CLINICAL TRIAL: NCT01547728
Title: Response of Recombinant Antithrombin in Heparin Resistant Patients Undergoing Cardiac Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Too many barriers to enroll participants.
Sponsor: Mayo Clinic (Other)
Collaborators: rEVO Biologics (Industry)
Responsible Party: Principal Investigator, William C. Oliver, Consulatant Cardio/Thoracic Anesthesia, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-004125
Record Dates: First submitted 2012-02-07; First posted 2012-03-08 (Estimated); Results first posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Thrombophilia Due to Acquired Antithrombin III Deficiency
Keywords: antithrombin; Heparin Resistant; Cardiac Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant antithrombin (rhAT) (Experimental): Subjects will receive an intravenous bolus of 500 units of recombinant, human antithrombin (rhAT, ATRYN ®). If the subject remains heparin-resistant, one more IV bolus of 500 units rhAT is given.
  Interventions: Drug: Recombinant antithrombin (rhAT)

INTERVENTIONS:
Drug: Recombinant antithrombin (rhAT) — Subjects will receive an intravenous bolus of 500 units of recombinant, human antithrombin (rhAT, ATRYN ®). If the subject remains heparin-resistant, one more IV bolus of 500 units rhAT is given.
  Other Names: ATryn®

SUMMARY:
The objective of this study is to prospectively evaluate the response of recombinant antithrombin (rAT) (ATRYN) in patients who are heparin resistant and are scheduled to undergo cardiac surgery.

DETAILED DESCRIPTION:
AT is an α2-globulin that is produced primarily in the liver. It binds thrombin, as well as other serine proteases, factors IX, X, XI, and XII, kallikrein, and plasmin irreversibly, which neutralizes their activity. However, only inhibition of thrombin and factor Xa by AT has physiologic and clinical significance.1 AT deficiency may occur as a congenital or acquired deficiency. Acquired deficiencies are secondary to increased AT consumption, loss of AT from the intravascular compartment (renal failure, nephrotic syndrome) or liver disease (cirrhosis). A normal AT level is 80% to 120% with activity below 50% considered clinically important based on the risk of venous thrombosis in patients with congenital deficiency of AT.2 However, the risk of thrombosis is higher in congenital forms than acquired forms of AT deficiency.3, 4 Unfortunately, the only abnormal coagulation test associated with this condition is the assay for AT activity, which is diagnostic but not readily available.

Acquired deficiencies of AT are commonly encountered in cardiac surgical patients. Anticoagulation with heparin for CPB depends on AT to inhibit clotting as heparin alone has no effect on coagulation. Heparin catalyzes AT inhibition of thrombin over a 1000 fold by binding to a lysine residue on AT and altering its conformation. Thrombin actually attacks AT, disabling it, but in the process attaches AT to thrombin, forming a complex that can be detected and used to assess thrombin formation but has no activity. Thirty percent of AT is consumed during this process so AT levels are reduced temporarily. If AT levels are not restored, then a condition may arise called heparin resistance. There are other less frequent causes of heparin resistance besides AT deficiency such as platelets, fibrin, vascular surfaces and plasma proteins.5 There is no universally accepted definition of heparin resistance. It is broadly defined as the failure of a specific heparin dose (300 - 400 u/kg) to prolong an ACT beyond 400 - 480 seconds in preparation for initiation of CPB. Because the definition of heparin resistance may differ according to both heparin dose and target ACT, the incidence of heparin resistance in the literature is very variable. A recent randomized prospective study analyzing 2270 cardiac cases, identified 3.7% of the patients to be heparin resistant but the incidence has been reported as high as 18% - 30% The incidence of heparin resistance is likely to further increase as the use of heparin infusions prior to cardiac surgery becomes more prevalent.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery requiring cardiopulmonary bypass (CPB)
* Heparin resistant according to this definition: initial activated clotting time (ACT) after an intravenous loading dose of heparin (300 u/kg) is less than 480 seconds

Exclusion criteria:

* current use of one or more of these medications:

  * warfarin (within 3 days of surgery);
  * streptokinase;
  * tissue plasminogen activator;
  * abciximab,
  * eptifibatide,
  * tirofiban or
  * clopidogrel.
* known hypersensitivity to goat or goat milk proteins,
* patients with pre-existing coagulopathy defined as a history of bleeding or laboratory bleeding disorder (e.g., von Willebrand disease, platelet disorder) and
* patients receiving direct thrombin inhibitors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Oliver, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Recombinant Antithrombin (rhAT)
Started | 42
Completed | 1
Not Completed | 41
Not completed — Change in procedure and equipment | 1
Not completed — Drug not ready for subject | 1
Not completed — Screen failure | 39

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Antithrombin (rhAT)
Number analyzed (Participants) | 42
Age, Continuous [Mean (Full Range); unit: years] | 64 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Whose Activated Clotting Time (ACT) is Prolonged Beyond 480 Seconds With Recombinant Human Antithrombin Concentrate (rhAT) Administration
Description: Restored antithrombin level is defined as an activated clotting time > 480 seconds 3 minutes after the initial dose of 500 units of rhAT is administered. The percentage of patients who meet this criterion will be summarized using a point estimate and a 95% confidence interval.
Time Frame: 3 minutes after the initial dose of rhAT, Day 1 of the study
Population: The study was terminated because there were too many barriers to enroll participants.
Arm/Group | Recombinant Antithrombin (rhAT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Recombinant Antithrombin (rhAT)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated because there were too many barriers to enroll participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days